CLINICAL TRIAL: NCT01791439
Title: Glossopharyngeal Nerve Blockade for Awake Videolaryngoscope Assisted Endotracheal Intubation in the Morbidly Obese.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Victoria Hospital, Canada (Other)
Responsible Party: Principal Investigator, Albert Moore, Dr., Royal Victoria Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 11-201-SDR; 11-201-SDR (Other: research ethics office)
Record Dates: First submitted 2013-02-10; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Gagging
MeSH Terms: conditions — Gagging | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Experimental): Patients in this arm will have gauze soaked with lidocaine applied to the peritonsillar pillars.
  Interventions: Other: lidocaine
- Saline (Placebo Comparator): Application of saline to the glossopharyngeal nerve.
  Interventions: Other: placebo

INTERVENTIONS:
Other: lidocaine — Application of lidocaine to the glossopharyngeal nerve.
  Arms: Lidocaine
Other: placebo
  Arms: Saline

SUMMARY:
The investigators wish to determine if application of 2% lidocaine soaked gauze to the peritonsillar pillars will decrease the amount of gagging caused by awake videolaryngocope assisted tracheal intubation in the morbidly obese.

ELIGIBILITY:
Inclusion Criteria:

* morbid obese patients scheduled for bariatric surgery, with a planned awake intubation.

Exclusion Criteria:

* inability to communicate in English or french
* allergies to any study drugs
* any patient with an American society of anesthesiologists score of 4 or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Gagging | 2 minutes
  We will assess the amount of gagging during the awake intubation.

SECONDARY OUTCOMES:
vital signs | 2 minutes
  we will asses vital signs during intubation.
lidocaine levels | 40 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada